CLINICAL TRIAL: NCT04984551
Title: ECHO Telementoring to Improve Quality Palliative Care in Underserved Areas of Kenya, Nigeria, Ghana, South Africa, India, and Ethiopia
Brief Title: Impact of Project ECHO on Improving the Quality of Palliative Care in Patients With Advanced Cancer and Their Caregivers in Underserved Areas of Kenya, Nigeria, Ghana, South Africa, India, and Ethiopia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-0462; NCI-2020-06074 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0462 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-08-27; First posted 2021-07-30 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm I: ECHO Participants (ECHO clinics, workshop, education) (Experimental): Participants participate in online ECHO clinics over 1 hour twice monthly for 12 months and in-country workshops twice per year. Participants also receive 5 core lectures through an internet-based professional education curriculum.
  Interventions: Other: Extension of Community Health (ECHO) Telementoring Clinic; Other: In-Country Workshops; Other: Professional Oncology Educations Programs
- Arm II: Patients (questionnaire, medical chart review) (Experimental): Patients complete 3 in-person or phone questionnaires over a total of 20 minutes every 3 months for 2 years about their symptoms, emotional and physical well-being, and their experience and satisfaction with outpatient oncology care. Patients' medical charts are reviewed for data collection. Patients complete a 15 minute interview in person or phone about the care they received by their physician at baseline, end of month 4 and month 12.
  Interventions: Other: Medical Chart Review; Other: Questionnaire Administration
- Arm III: Caregivers (questionnaire) (Experimental): Caregivers complete an in-person or phone questionnaire over 5 minutes up to 8 times about their experience and satisfaction with the cancer care their family member has received. Caregivers complete a 15-minute interview in person or by phone their family member received by their physician.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Other: Extension of Community Health (ECHO) Telementoring Clinic — Participate in ECHO clinics presenting cases for guidance and feedback
  Arms: Arm I: ECHO Participants (ECHO clinics, workshop, education)
Other: In-Country Workshops — In-Country Workshops Participate in hands-on training and workshops
  Arms: Arm I: ECHO Participants (ECHO clinics, workshop, education)
Other: Professional Oncology Educations Programs — Receive 5 core online lectures
  Arms: Arm I: ECHO Participants (ECHO clinics, workshop, education)
Other: Medical Chart Review — Medical charts are reviewed for data collection
  Other Names: Chart Review
  Arms: Arm II: Patients (questionnaire, medical chart review)
Other: Questionnaire Administration — Complete questionnaire(s)
  Arms: Arm II: Patients (questionnaire, medical chart review); Arm III: Caregivers (questionnaire)

SUMMARY:
This trial investigates the experience and satisfaction of care in patients with cancer that has spread to other places in the body (advanced) and their caregivers living in underserved areas of Kenya, Nigeria, Ghana, South Africa, India and Ethiopia as part of Project Extension for Community Healthcare Outcomes (ECHO). Project ECHO is a model of medical education and care management that empowers clinicians to provide better care to more people where they live. Understanding the experiences and satisfaction of patients and caregivers may help improve healthcare workforce capacity and increase access to specialty care for the world's rural and underserved populations.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effects of Project ECHO on patient-reported quality of life (QOL) (as assessed by the change in Functional Assessment of Cancer Illness Therapy FACT-General [G]) in seriously ill patients of providers receiving ECHO model-based comprehensive educational and telementoring intervention (ECHO-Palliative Care, or ECHO-PCT).

SECONDARY/EXPLORATORY OBJECTIVES:

I. To examine the effects of ECHO-PCT on patients' symptom distress as assessed by the Edmonton Symptom Assessment Scale (ESAS), Symptom Distress Scores (SDS), as well as patient and caregiver experience and satisfaction as assessed by the FAMCARE-P 16-item (16)-patient and FAMCARE-caregiver questionnaires.

II. To explore the effects of ECHO-PCT on providers' efficacy in, knowledge of, and competence to deliver Palliative Care to Patients with serious life limiting illness, as well as their satisfaction with providing Palliative Care services as assessed by Palliative Care Participant Initial Survey, Palliative Care Participant Follow Up Survey, and Feedback Survey.

IIa. Increase patient access to quality palliative care in these regions (morphine consumption).

IIb. Increase patient access to quality palliative care in these regions (morphine consumption).

IIc. Increased patient access to palliative care (PC) measured by the number of patient visits (new and follow-ups).

IId. Provider turnover. IIe. Adherence, measured by the number of ECHO sessions held, the number of ECHO participants at each session, and the number of cases reviewed.

IIf. Comfort with the ECHO platform and ability to learn/engage via distance technology, assessed by the Palliative Care Participant Initial Survey and Palliative Care Participant Follow Up Survey.

OUTLINE: Participants are assigned to 1 of 3 arms.

ARM I (ECHO PARTICIPANTS): Participants participate in online ECHO clinics over 1 hour twice monthly for 12 months and in-country workshops twice per year. Participants complete 5 online surveys between baseline through end of year 2 for up to a total of 26 minutes .Participants complete a 15-minute interview in person or phone about their experience in the ECHO project.

ARM II (PATIENTS): Patients complete 3 in-person or phone questionnaires over a total of 20 minutes every 3 months for 2 years about their symptoms, emotional and physical well-being, and their experience and satisfaction with outpatient oncology care. Patients' medical charts are reviewed for data collection. Patients complete a 15-minute interview in person or phone about their care received by their physician at baseline, end of month 4 and month 12.

ARM III (CAREGIVERS): Caregivers complete an in-person or phone questionnaire over 5 minutes up to 8 times about their experience and satisfaction with the cancer care their family member has received. Caregivers complete a 15 minute interview in person or by phone about the care their family member received by their physician.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT: Scheduled to receive treatment at participating primary care practice for advanced cancer
* PATIENT: 18 years or older
* PATIENT: Willing to be accessible to the research team for follow-up by telephone or in person
* PATIENT: Prognosis of at least 1 year as ascertained by the treating physician
* PATIENT: Able to read and understand English as assessed by the treating physician
* CAREGIVER: Identified or self-identified as primary caregiver of the patient
* CAREGIVER: Willing to be accessible to the research team for follow-up by telephone or in person
* CAREGIVER: 18 years or older
* CAREGIVER: Able to read and understand English as assessed by the treating physician
* ECHO PARTICIPANT: Participant must be a health care provider interested to participate in the study for 2 years and understand the protocol and provide consent
* ECHO PARTICIPANT: Able to read and understand English as assessed by principal investigator (PI)

Exclusion Criteria:

* Unable to understand and sign consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in patients' quality of life | Baseline up to 12 months
  Measured by Functional Assessment of Cancer Illness Therapy FACT-General (FACT-G). A 27-item compilation of general questions divided into four primary domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being. Each question is assessed using a Likert scale ranging from 0 to 4. The FACT-G total score is the sum of the domain scores..

SECONDARY OUTCOMES:
Change in patients' symptom distress | Baseline up to 2 years
  Will be assessed by the Edmonton Symptom Assessment Scale, Symptom Distress Scores, (ESAS-SDS). The ESAS is a validated questionnaire measuring 10 symptoms (pain, fatigue, nausea, depression, anxiety, drowsiness, shortness of breath, appetite, sleep, and well-being). It has good reliability and can be completed within minutes. The ESAS-SDS will be calculated by the sum of the symptom scores of measures ESAS Pain, ESAS Fatigue, ESAS nausea, ESAS Depression, ESAS anxiety, ESAS drowsiness, ESAS Dyspnea, ESAS Appetite, ESAS Well-being.
Patients' satisfaction of care | Baseline up to 2 years.
  Assessed by FAMCARE P16, a self-report scale assessing patient experience and satisfaction with outpatient palliative oncology care, which is composed of 16 items rated from 1 (very dissatisfied) to 5 (very satisfied). The items are not specific for a particular tumor type or symptom but are broadly relevant for outpatients with advanced cancer; the summed items produce a single satisfaction score.
Caregivers' satisfaction of care | Baseline up to 2 years
  Assessed by FAMCARE -cg scale, which measures the degree of experience and satisfaction of the caregivers with health care in terms of information provided, availability of care, physical individual with advanced cancer care, and psychological care for patients.
Providers' efficacy in knowledge of delivering palliative care | Baseline
  Assessed by completing the Palliative Care Participant Initial Survey
Providers' efficacy in knowledge of delivering palliative care | Up to 2 years
  Assessed by completing the Palliative Care Participant Follow up Survey composed of 9 questions about providers' knowledge of assessments performed in the palliative care setting.
Providers' competence to deliver palliative care | Baseline up to 2 years
  Measured by the distance technology sessions held twice monthly.
Providers' Satisfaction and feedback | Baseline up to 2 years
  Assessed by completing 7 questions about providers' opinions of distance learning technology.
Burnout among ECHO participant | Baseline up to 2 years
  Measured by Maslach Burnout Inventory-Human Services Survey (MBI-HSS). It consists of three factors (depersonalization [DP], emotional exhaustion [EE], and personal achievement [PA]) with 22 items, each scored on a 7-point Likert scale. DP and EE scores are positively correlated with burnout, while PA is negatively correlated.

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org